CLINICAL TRIAL: NCT05820906
Title: Cadonilimab Plus Regorafenib and Gem-Cis Chemotherapy in Advanced Biliary Tract Cancer: A Single Center, Single Arm, Phase II Trial
Brief Title: Cadonilimab Plus Regorafenib and Gem-Cis Chemotherapy in Advanced Biliary Tract Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, HuiKai Li, Professor and Chief Surgeon, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-C-N1-0057
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Advanced Biliary Tract Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab+rego+Gem/Cis (Experimental)
  Interventions: Drug: Cadonilimab+Regorafenib+GC

INTERVENTIONS:
Drug: Cadonilimab+Regorafenib+GC — Cadonilimab:10mg/kg, iv,q3w,D1 Regorafenib: 80mg, po, orally once daily Gemcitabine:1000 mg/m2, iv, Q3W，D1,D8 Cisplatin:25 mg/m2, iv, Q3W, D1,D8

SUMMARY:
To evaluate the efficacy and safety of Cadonilimab in combination with Regorafenib and Gem-Cis chemotherapy in advanced biliary tract Cancer

ELIGIBILITY:
Main Inclusion Criteria:

1. subjects with a histopathological or cytologically diagnosis of BTC
2. The participants must be required to sign an informed consent
3. At least one measurable lesion (RECIST 1.1)
4. No previous systematic treatment for BTC
5. Child-Pugh Score, Class A
6. ECOG performance status 0 or 1
7. Adequate organ function
8. Life expectancy of at least 3 months

Exclusion Criteria:

1. Diagnosis of mixed ampullary, hepatocellular and cholangiocarcinoma
2. Known history of serious allergy to any monoclonal antibody
3. Known central nervous system metastases and/or leptomeningeal disease prior to treatment
4. Portal hypertension with esophageal or gastric varices within 6 months prior to initiation of treatment
5. Any bleeding or thrombotic disorder within 6 months prior to initiation of treatment
6. Any active malignancy prior to the start of treatment
7. Active or history of autoimmune disease
8. Other acute or chronic conditions, psychiatric disorders, or laboratory abnormalities that may increase the risk of study participation
9. Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate ( ORR) per RECIST 1.1 | Up to 1 year
  Defined as proportion of patients who have a best response of CR or PR

SECONDARY OUTCOMES:
Overall survival (OS) | Up to two years
  Defined as the time from enrollment to death from any cause
Progress Free Survival (PFS) | Up to two years
  Defined as the time from enrollment to disease progression or death (whichever occurs first)
Adverse Events (AEs) | Up to two years
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0
Disease control rate (DCR) per RECIST 1.1 | Up to 1 year
  Defined as proportion of patients who have CR or PR or SD

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No